CLINICAL TRIAL: NCT04105153
Title: Real-world Analysis of Workup at Disease Progression and Implementation of Osimertinib for EGFR+ NSCLC
Status: Completed | Type: Observational
Sponsor: Thoraxklinik-Heidelberg gGmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: S-469/19; ESR-19-14460 (Other: AstraZeneca)
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer
Keywords: Non-small cell lung carcinoma; EGFR mutation; Tyrosine Kinase Inhibitor; Osimertinib; EGFR T790M
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TKI-treated advanced EGFR+ NSCLC: Patients with advanced EGFR-mutated non-small cell lung cancer treated with tyrosine kinase inhibitors

SUMMARY:
Tyrosine kinase inhibitors (TKI) have greatly improved prognosis of epidermal growth factor receptor (EGFR)-positive non-small cell lung cancer (NSCLC), with tumor responses in the majority of cases and a median overall survival currently exceeding 2.5 years. However, clinical courses vary widely and eventual treatment failure is inevitable. The most common resistance mechanism against first- and second-generation EGFR inhibitors is the EGFR T790M mutation, which emerges in about 50% of cases and is amenable to next-line treatment with the third-generation compound osimertinib. However, experience in everyday clinical practice shows that implementation of EGFR TKI sequencing is often problematic, for example because a considerable number of EGFR+ NSCLC patients failing first- and second-generation EGFR inhibitors do not undergo T790M mutation testing at the time of disease progression. This study will use patient records to analyze the clinical course of EGFR+ NSCLC patients treated with first- and second-generation EGFR inhibitors at the Thoraxklinik Heidelberg (Germany) during the past years. The main aim is to analyze the diagnostic and therapeutic measures, including implementation of osimertinib, taken at the time of disease progression as well as their effect on patient outcome in a real-world, routine clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed locally advanced (stage III) and not suitable for definitive local treatment, or metastatic (stage IV) NSCLC
* activating EGFR mutation confirmed
* treatment with EGFR TKI

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All NSCLC patients with activating EGFR mutations treated with EGFR TKI at the Thoraxklinik Heidelberg between 2010 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Fraction of EGFR+ NSCLC patients with sequential TKI treatment | assessment will performed retrospectively for all study patients from September 2019 until June 2020
  * the rate of rebiopsy and molecular workup (especially T790M testing) at disease progression under treatment with first-/second-generation EGFR inhibitors
  * the frequency of T790M mutations in the molecular workup of patients with disease progression under first-/second-generation EGFR inhibitors
  * the actual rate of osimertinib implementation after failure of first-/second-generation EGFR inhibitors in the "real-world" setting.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | assessment will performed retrospectively for all study patients from September 2019 until June 2020
  Progression-free survival (PFS) of patients treated with first-/second-generation EGFR inhibitors and/or osimertinib in the real-world setting
Time-to-next-treatment (TNT) | assessment will performed retrospectively for all study patients from September 2019 until June 2020
  Time-to-next-treatment (TNT) of patients treated with first-/second-generation EGFR inhibitors and/or osimertinib in the real-world setting
Time-to-chemotherapy (TTC) | assessment will performed retrospectively for all study patients from September 2019 until June 2020
  Time-to-chemotherapy (TTC) of patients treated with first-/second-generation EGFR inhibitors and/or osimertinib in the real-world setting
Overall survival (OS) | assessment will performed retrospectively for all study patients from September 2019 until June 2020
  Overall survival (OS) of patients treated with first-/second-generation EGFR inhibitors and/or osimertinib in the real-world setting

CONTACTS AND LOCATIONS:
Overall Officials: Petros Christopoulos, MD, Principal Investigator — Thoraxklinik Heidelberg gGmbH - Universitätsklinikum Heidelberg
Locations (1):
- Thoraxklinik-Heidelberg gGmbH - Universitätsklinikum Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Background] Schrank Z, Chhabra G, Lin L, Iderzorig T, Osude C, Khan N, Kuckovic A, Singh S, Miller RJ, Puri N. Current Molecular-Targeted Therapies in NSCLC and Their Mechanism of Resistance. Cancers (Basel). 2018 Jul 4;10(7):224. doi: 10.3390/cancers10070224. PMID 29973561
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926